CLINICAL TRIAL: NCT03805100
Title: A Phase III Double-Blind, Parallel Group, Multicenter Study to Compare the Efficacy and Safety of Xlucane Versus Lucentis® in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Comparing the Efficacy and Safety of Biosimilar Candidate Xlucane Versus Lucentis® in Patients With nAMD
Acronym: XPLORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xbrane Biopharma AB (Industry)
Collaborators: Stada Arzneimittel AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XBR1001
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-02

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xlucane (Experimental): Xlucane (0.05 mL of 10 mg/mL ranibizumab) in the study eye monthly for 52 weeks.
  Interventions: Biological: Ranibizumab
- Lucentis (Active Comparator): Lucentis (0.05 mL of 10 mg/mL ranibizumab) in the study eye monthly for 52 weeks.
  Interventions: Biological: Ranibizumab

INTERVENTIONS:
Biological: Ranibizumab — Intravitreal injection

SUMMARY:
The objectives of the study are to demonstrate the equivalence of Xlucane to Lucentis® in treatment of subjects with wet (ie, neovascular) age-related macular degeneration (wAMD).

DETAILED DESCRIPTION:
This is a phase III multicenter, double-masked, randomized, parallel group study in subjects with wAMD. Approximately 580 subjects will be enrolled and randomized in a 1:1 ratio to receive either Lucentis® or the investigational product, Xlucane in the study eye once every 4 weeks for 52 weeks. The study eye will be defined as the eye meeting the enrollment criteria. The assigned study drug will be administered as an ophthalmic intravitreal (IVT) injection. A subgroup of 60 subjects at a select number of participating sites will be sequentially asked to participate in an evaluation of PK.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent form obtained at screening, before any study-related procedures.
* Willingness and ability to undertake all scheduled visits and assessments as judged by the investigator.
* Newly diagnosed, active subfoveal Choroidal Neovascularization (CNV) lesion secondary to age-related macular degeneration (AMD) in the study eye. Note: Active CNV indicates the presence of leakage as evidenced by Fluorescein Angiography (FA) and intra- or subretinal fluid as evidenced by Optical Coherence Tomography (OCT) which must be confirmed by the central reading center during Screening:

  1. The area of CNV must be ≥ 50% of the total lesion area in the study eye, and
  2. Total lesion area ≤ 9.0 Disc Areas (DA) in size (including blood, scars and neovascularization) as assessed by FA in the study eye.
* Best Corrected Visual Acuity (BCVA) of ≤ 73 and ≥ 49 ETDRS letter score in the study eye, using ETDRS chart (20/40 to 20/100 Snellen equivalent) at Screening.
* Fellow eye should not be expected to need any anti-VEGF treatment for the duration of study participation.
* Age ≥ 50 years at screening.
* Male and female subjects of childbearing potential must be willing to completely abstain or agree to use an appropriate method of contraception, from the time of signing informed consent and for the duration of study participation through 3 months, following the last dose of study drug.

Exclusion Criteria:

* Any previous intervention including pharmacological treatment, laser and/or surgery for wAMD in either eye; (Exception: Vitamin supplementation for AMD prevention).
* Any previous vitreoretinal surgery in the study eye for any cause.
* Any previous IVT treatment including any anti-VEGF medications, steroids and/or any other investigational medication in either eye.
* The use of long-acting steroids, either systemic or intraocular in any eye, in the 18 months before planned initiation of study treatment. (Note: Iluvien® [fluocinolone acetonide intravitreal], current or planned implantation during the study, is prohibited.)
* Subfoveal fibrosis, atrophy or scarring extending > 50% of total lesion area, in the study eye as assessed by the investigator at screening and confirmed by the central reading center prior to randomization.
* Choroidal neovascularization in either eye due to non-AMD causes (eg, DME, RVO, ocular histoplasmosis or trauma, etc.) as assessed by FA and confirmed by central reading center.
* Active or recent (within 28 days prior to randomization) intraocular, extraocular, and periocular inflammation or infection in either eye.
* History of idiopathic or autoimmune-associated uveitis in either eye.
* Infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye.
* Unmedicated intraocular pressure (IOP) ≥ 30 mmHg at Screening in either eye.
* Topical ocular corticosteroids administered for ≥ 30 consecutive days in the study eye within 90 days prior to Screening.
* Spherical equivalent of the refractive error in the study eye demonstrating more than 8 diopters of myopia.
* Corneal transplant or corneal dystrophy in the study eye.
* History of rhegmatogenous retinal detachment in the study eye.
* History of macular hole in the study eye.
* Retinal pigment epithelial tear or rip, involving the macula in the study eye as assessed by FA and confirmed by the central reading center.
* Current vitreous hemorrhage in the study eye.
* Subretinal hemorrhage that is ≥ 50% of the total lesion area in the study eye, or if the subretinal hemorrhage involves the fovea is 1 or more DA (≥ 2.54 mm2) in size in the study eye, as assessed by FA and confirmed by the central reading center.
* Other intraocular surgery (including cataract surgery) in the study eye within the 3 months prior to baseline. The yttrium aluminum garnet [YAG] posterior capsulotomy is allowed not later than 4 weeks prior to screening.
* Any concurrent intraocular condition in the study eye (eg, cataract or diabetic retinopathy) that, in the opinion of the investigator, could require treatment during the study period to prevent or treat loss of visual acuity.
* Significant media opacities (including cataract) in the study eye interfering with BCVA assessment or fundus imaging (FA/FP/OCT).
* Aphakia or absence of the posterior capsule in the study eye, unless it occurred as a result of a YAG posterior capsulotomy in association with prior posterior chamber intraocular lens implantation.
* Presence of advanced glaucoma or optic neuropathy that involve(s) or threaten(s) the central visual field in the study eye (as judged by the investigator).
* History of glaucoma filtering surgery or argon laser trabeculoplasty in the study eye (Exception: Laser iridotomy and selective laser trabeculoplasty are allowed).
* Uncontrolled ocular glaucoma or hypertension in the study eye, defined as IOP ≥ 25 mmHg despite treatment with anti-glaucoma medication.
* Any previous systemic anti-VEGF treatment (eg, bevacizumab).
* Contraindication for Lucentis® (hypersensitivity to ranibizumab or to any of the study treatment excipients).
* Current treatment for active systemic infection.
* Females who are pregnant, nursing, planning a pregnancy during the study, or of childbearing potential and not using a reliable method of contraception and/or not willing to use a reliable method of contraception during their participation in the study.
* Participation in another clinical trial within the previous 3 months or any other clinical trial of anti-angiogenic drugs.
* Reasonable suspicion of other disease or condition that might render the subject at a high risk of treatment complications or otherwise confound interpretation of the study results (as judged by the investigator).
* PK subgroup only: Contraindication for additional blood sampling (as judged by the investigator).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anat Loewenstein, Professor, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (102):
- United States (26):
  - Retinal Research Institute, LLC, Gilbert, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Centers P.C, Tucson, Arizona
  - Win Retina, Arcadia, California
  - The Retina Partners, Encino, California
  - Mark B. Kislinger MD Inc., Glendora, California
  - Retina Consultants Medical Group Inc., Sacramento, California
  - Colorado Retina Associates, Golden, Colorado
  - Fort Lauderdale Eye Institute, Fort Lauderdale, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, Marietta, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - Sabates Eye Centers, Leawood, Kansas
  - Retina Vitreous Surgeons of Central New York PC, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Houston Eye Associates, Houston, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group LLC, Willow Park, Texas
- Bulgaria (5):
  - Specialized Eye hospital for active treatment Luxor, Plovdiv
  - Specialized eye clinic Zrenie, Sofia
  - Specialized Eye hospital for active treatment Acad. Pashev, Sofia
  - Specialized Hospital for Active Treatment of Eye Diseases "Zora", Sofia
  - AMCSMP Eye Clinic St. Petka, Varna
- Czechia (5):
  - Všeobecná FN v Praze, Brno
  - Oční klinika, Fakultní nemocnice, Hradec Králové
  - Faculty Hospital Kralovske Vinohrady, Prague
  - VFN Ocni klinika, Prague
  - Axon-Clinical, s.r.o., Prague
- Estonia (2):
  - OÜ Dr Kai Noor Silmakabinet, Tallinn
  - Mustame Eye Centre, Tallinn
- Hungary (11):
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Department of Ophthalmology, Semmelweis University, Budapest
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Szent Imre Teaching Hospital, Budapest
  - Budapest Retina Associates, Budapest
  - Jahn Ferenc South-Budapest Hospital, Budapest
  - University of Debrecen, Debrecen
  - Szabolcs-Szatmr-Bereg County Hospital, Nyíregyháza
  - Ganglion Medical Center, Pécs
  - Markusovszky University Teaching Hospital, Szombathely
  - Zalan Megyei Szent Rafael kórház, Zalaegerszeg
- Rising Retina Clinic, Ahmedabad, India
- Israel (11):
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Tel Aviv Sourasky Medical Centre, Tel Aviv
  - Asaf Harofe Hospital, Zrifin
- Latvia (2):
  - P.Stradins University Hospital, Riga
  - The Dr Solomatin Eye Center, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (6):
  - Klinika Okulistyczna Oftalmika, Bydgoszcz
  - Professor K. Gibinski University Clinical Centre, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - Dr Nowosielska Okulistyka i Chirurgia Oka, Warsaw
  - Retina Okulistyka Sp. z o.o. sp. km, Warsaw
- Romania (2):
  - Clinica Retina, Bucharest
  - Opticlass Timisoara, Timișoara
- Russia (6):
  - FGAU NMRC MNTK Eye Microsurgery n.a. acad. S.N. Fyodorov Cheboksary Branch, Cheboksary
  - LLC Kuzlyar, Kazan'
  - Federal State Budget Scientific Institute of Eye Diseases, Moscow
  - S. Fyodorov Eye Microsurgery Federal State Institution, Moscow
  - S.Fyodorov Eye Microsurgery Federal State Institution, Saint Petersburg
  - First Pavlov State Medical University of St.Petersburg, Saint Petersburg
- Slovakia (4):
  - F.D.Roosevelt Hospital, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Fakultna nemocnica Trencin, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- Spain (14):
  - Hospital General Universitario de Albacete, Albacete
  - Instituto de Microcirugia Ocular, Barcelona
  - Hospital de Viladecans, Barcelona
  - Bellvitge University Hospital, L'Hospitalet de Llobregat
  - Hospital Universitario Puerta de Hierro-Majadahonda, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Clinica Universidad de Navarr, Pamplona
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen Macarena, Seville
  - Unit of Macula. Oftalvist Clinic, Valencia
  - FISABIO-Oftalmologia Medica FOM, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Ukraine (5):
  - Regional Clinical Hospital Center for Emergency Medical Care And Disaster Medicine, Kharkiv
  - Medical and Diagnostic Centre PE PMC "Acinus", Kropyvnytskyi
  - Filatov Institute of Eye Diseases Tissue Therapy, Odesa
  - Clinic of Professor Serhiienko, Vinnitsa
  - Medical center LTD VISUS, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Xlucane (Proposed Ranibizumab Biosimilar): Xlucane (proposed ranibizumab biosimilar) in the study eye monthly for 52 weeks by intravitreal injection.
- Lucentis (Ranibizumab): Lucentis (ranibizumab) in the study eye monthly for 52 weeks by intravitreal injection
Period: Overall Study
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Started | 292 (Number of participants randomized to Xlucane.) | 290 (Number of participants randomized to Lucentis.)
Completed | 245 (Number of participants completing the treatment per protocol.) | 241 (Number of participants completing the treatment per protocol.)
Not Completed | 47 | 49

BASELINE CHARACTERISTICS:
Population: All 292 subjects in the Xlucane group, and 289 out of the 290 subjects in the Lucentis group were dosed with study drug. 1 subject in the Lucentis group withdrew consent after randomization, and was never treated, therefore was never exposed to study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab) | Total
Number analyzed (Participants) | 292 | 290 | 582
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 32 | 66
  >=65 years | 258 | 258 | 516
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.5 (8.68) | 73.8 (8.25) | 74.1 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 157 | 325
  Male | 124 | 133 | 257
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 44 | 42 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 248 | 248 | 496
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: Letters] | 61.7 (8.11) | 61.5 (8.20) | 61.6 (8.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: Change(s) in BCVA letters at Week 8 compared to baseline using the ETDRS protocol
Time Frame: Baseline and Week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Letters
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
Letters | 4.57 [3.54 to 5.61] | 6.37 [5.31 to 7.42]

2. Secondary Outcome: Change From Baseline in the Total Size of Choroidal Neovascular Leakage Area in the Study Eye
Description: Change in the total size of choroidal neovascular leakage area in the study eye week 52 compared to baseline measured by Fluorescein Angiography
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mm2
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
mm2 | -4.09 [-4.66 to -3.52] | -3.71 [-4.28 to -3.14]

3. Secondary Outcome: Change From Baseline in the Total Size of Choroidal Neovascularisation in the Study Eye
Description: Change From Baseline in the Total Size of Choroidal Neovascularisation in the Study Eye Measured by Fluorescein Angiography
Time Frame: Baseline and week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: mm2
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
mm2 | -1.62 [-2.19 to -1.05] | -1.11 [-1.68 to -0.54]

4. Secondary Outcome: Central Foveal Thickness in the Study Eye
Description: Central Foveal Thickness in the Study Eye Measured by Optical Coherence Tomography
Time Frame: Baseline to week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
um | -117.44 [-125.33 to 109.55] | -115.14 [-123.14 to -107.14]

5. Secondary Outcome: Percentage of Subjects With Loss of <15 BCVA Letters
Description: Percentage of Subjects With Loss of <15 BCVA Letters Compared to Baseline in the Study Eye
Time Frame: Baseline to week 52
Measure: Number; unit: percentage of responders
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
percentage of responders
  Missing at random (MAR) | 94.8 | 96.0
  Missing completely at random (MCAR) | 94.9 | 96.1
  Missing not at random (MNAR) | 94.8 | 96.1
  Composite (Missing and non-evaluable data are classed as no response) | 68.8 | 67.6

6. Secondary Outcome: Percentage of Subjects With Gain of ≥15 BCVA Letters
Description: Percentage of Subjects With Gain of ≥15 BCVA Letters Compared to Baseline in the Study Eye
Time Frame: Baseline to week 52
Measure: Number; unit: percentage of responders
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
percentage of responders
  Missing at random (MAR) | 23.6 | 29.7
  Missing completely at random (MCAR) | 23.2 | 28.8
  Missing not at random (MNAR) | 23.6 | 30.4
  Composite (Missing and non-evaluable data are classed as no response) | 17.1 | 21.4

7. Secondary Outcome: Subretinal Fluid in the Study Eye
Description: Change from Baseline in the Amount of Subretinal Fluid in the Study Eye Measured by OCT
Time Frame: Baseline to week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
um | -34.88 [-39.07 to -30.69] | -32.93 [-37.21 to -28.65]

8. Secondary Outcome: Width of Retinal Pigment Epithelium Detachments in the Study Eye
Description: Change from Baseline in the Width of Retinal Pigment Epithelium Detachments in the Study Eye Measured by OCT
Time Frame: Baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
um | -161.39 [-387.16 to -135.62] | -256.33 [-384.56 to -128.10]

9. Secondary Outcome: Pharmacokinetic Plasma Ranibizumab Concentrations
Description: Pharmacokinetic Plasma Ranibizumab Concentrations (sub-study)
Time Frame: Day 1 to week 20
Population: 70 patients were included in the PK substudy
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 40 | 30
pg/mL
  Day 1 | 2230 (1429) | 2190 (1336)
  Week 20 | 2450 (1384) | 2150 (1233)

10. Secondary Outcome: Height of Retinal Pigment Epithelium Detachments
Description: Change from Baseline in the Height of Retinal Pigment Epithelium Detachments in the Study Eye Measured by OCT
Time Frame: Baseline to Week 52
Measure: Least Squares Mean (95% Confidence Interval); unit: um
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 292 | 290
um | -81.49 [-96.33 to -66.66] | -73.15 [-88.35 to -57.95]

ADVERSE EVENTS:
Time Frame: From the time the participant signed the written informed consent to 28 days [± 5 days] of receiving last dose of study drug, up to 53 weeks.
Description: AEs (ocular or non-ocular) as well as injection site reactions were recorded.
Arm/Group | Xlucane (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
All-Cause Mortality (participants affected / at risk) | 8/292 | 3/290
Serious Adverse Events (participants affected / at risk) | 33/292 | 35/290
Other Adverse Events (participants affected / at risk) | 25/292 | 33/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xlucane (Proposed Ranibizumab Biosimilar) (N=292) | Lucentis (Ranibizumab) (N=290)
Retinal pigment epithelial tear (Eye disorders) | 2 (2) | 1 (2)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Macular vasospasm (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Appendiceal Abscess (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Artrial fibrilation (Cardiac disorders) | 3 (3) | 2 (2)
Myocardial infraction (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkins disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulva cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xlucane (Proposed Ranibizumab Biosimilar) (N=292) | Lucentis (Ranibizumab) (N=290)
Conjunctival Haemorrhage (Eye disorders) | 15 (19) | 16 (22)
Hypertension (Vascular disorders) | 10 (10) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03805100/Prot_SAP_000.pdf